CLINICAL TRIAL: NCT01723800
Title: Phase I Trial of BKM120 in Combination With Carboplatin and Pemetrexed in Patients With Advanced Non-Squamous Non-Small Cell Lung Cancer (NSCLC)
Brief Title: PI3K Inhibitor BKM120, Carboplatin, and Pemetrexed Disodium in Treating Patients With Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12219; NCI-2012-02161 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — NVP-BKM120; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (pemetrexed, carboplatin, PI3K inhibitor BKM120) (Experimental): Patients receive pemetrexed disodium IV over 10 minutes followed by carboplatin IV over 30 minutes on day 1, and PI3K inhibitor BKM120 PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients may receive courses of PI3K inhibitor BKM120 alone or PI3K inhibitor BKM120 and pemetrexed disodium after 4-6 courses with carboplatin in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: PI3K inhibitor BKM120; Drug: pemetrexed disodium; Drug: carboplatin; Other: laboratory biomarker analysis; Other: pharmacological study; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: PI3K inhibitor BKM120 — Given PO
  Other Names: BKM120; PI3K_Inhibitor_BKM120; Buparlisib
Drug: pemetrexed disodium — Given IV
  Other Names: ALIMTA; LY231514; MTA
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This phase I trial studies the side effects and best dose of PI3K inhibitor BKM120 when given together with carboplatin and pemetrexed disodium in treating patients with stage IV non-small cell lung cancer. PI3K inhibitor BKM120 and pemetrexed disodium may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving PI3K inhibitor BKM120, carboplatin, and pemetrexed disodium together may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase 2 dose (RP2D) of BKM120 (PI3K inhibitor BKM120) that can be administered in combination with carboplatin and pemetrexed (pemetrexed disodium) in patients with advanced non-squamous non-small cell lung cancer (NSCLC).

II. To define the dose-limiting toxicity (DLT) and other toxicities associated with the use of combination BKM120 and carboplatin and pemetrexed.

SECONDARY OBJECTIVES:

I. To evaluate the pharmacokinetic parameters of BKM120, when used in combination with carboplatin and pemetrexed.

II. To obtain preliminary evidence of anti-tumor activity with this combination.

III. To evaluate downstream inhibition of the phosphatidylinositol 3 kinase (PI3K) pathway.

OUTLINE: This is a dose-escalation study of PI3K inhibitor BKM120. Patients receive pemetrexed disodium intravenously (IV) over 10 minutes followed by carboplatin IV over 30 minutes on day 1, and PI3K inhibitor BKM120 orally (PO) once daily (QD) on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients may receive courses of PI3K inhibitor BKM120 alone or PI3K inhibitor BKM120 and pemetrexed disodium after 4-6 courses with carboplatin in the absence of unacceptable toxicity or disease progression.

After completion of study treatment, patients are followed up for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have signed a written informed consent
* Patients must have a histologic or cytologic diagnosis of advanced, nonsquamous NSCLC (stage IV by American Joint Committee on Cancer [AJCC] 7th edition [ed.])
* Patients should not have received prior systemic chemotherapy for metastatic disease (prior epidermal growth factor receptor [EGFR], anaplastic lymphoma kinase [ALK], kinase inhibitor therapy is allowed); prior adjuvant or neoadjuvant therapy for early stage disease is allowed if received >= 12 months prior to study entry
* Prior radiation therapy is allowed to < 25% of the bone marrow; prior radiation must be completed at least 2 weeks prior to day 1 of cycle 1, and patients must have recovered from the acute toxic effects
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patients must have at least one site of measurable disease (per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin (Hb) > 9 g/dL
* Total calcium (corrected for serum albumin) within normal limits (bisphosphonate use for malignant hypercalcemia control is not allowed)
* Magnesium >= the lower limit of normal (LLN)
* Potassium within normal limits for the institution
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within normal range (or =< 3 x upper limit of normal [ULN] if liver metastases are present)
* Serum bilirubin within normal range (or =< 1.5 x ULN if liver metastases are present)
* Serum creatinine =< 1.5 x ULN or calculated or 24-hour clearance >= 45 mL/min (calculated creatinine clearance based on Cockcroft-Gault formula)
* Serum phosphorus >= LLN
* Serum amylase =< ULN
* Serum lipase =< ULN
* Fasting plasma glucose =< 120 mg/dL (6.7 mmol/L)
* Negative serum pregnancy test within 72 hours before starting study treatment in women with childbearing potential
* International normalized ratio (INR) =< 2

Exclusion Criteria:

* Patients who have received prior treatment with a P13K inhibitor or mammalian target of rapamycin (mTOR)-directed inhibitor
* Patients with a known hypersensitivity of BKM120 or to its excipients
* Patients with anaplastic lymphoma kinase (ALK) rearrangement or an activating epidermal growth factor receptor (EGFR) mutation who have not received and progressed on appropriate tyrosine kinase inhibitor therapy
* Patients with untreated brain metastases are excluded; however, patients with metastatic central nervous system (CNS) tumors may participate in this trial, if the patient is > 2 weeks from therapy completion (incl. radiation and/or surgery), is clinically stable at the time of study entry; stable corticosteroids treatment (e.g. dexamethasone 2 mg/day, prednisolone 10 mg/day) is permitted if it was initiated at least 14 days before start of study treatment
* Patients with acute or chronic liver, renal disease or pancreatitis
* Patient has any of the following mood disorders as judged by the investigator or a psychiatrist, or as a result of the patient's mood assessment questionnaire:

  * Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others) or patients with active severe personality disorders (defined according to Diagnostic and Statistical Manual of Mental Disorders [DSM]-IV) are not eligible; NOTE: for patients with psychotropic treatments ongoing at baseline, the dose and the schedule should not be modified within the previous 6 weeks prior to start of study drug
  * >= Common Terminology Criteria for Adverse Events (CTCAE) grade 3 anxiety
  * Meets the cut-off score of >= 10 in the Patient Health Questionnaire (PHQ)-9 or a cut-off of >= 15 in the Generalized Anxiety Disorder 7-item (GAD-7) mood scale, respectively, or selects a positive response of "1, 2, or 3" to question number 9 regarding potential for suicidal thoughts in the PHQ-9 (independent of the total score of the PHQ-9)
* Patients with diarrhea >= CTCAE grade 2
* Left ventricular ejection fraction (LVEF) < 50% as determined by echocardiogram (ECHO)
* Corrected QT interval (QTc) > 480 msec on screening electrocardiogram (ECG) (using the Fridericia correction QTc [QTcF] formula)
* Angina pectoris that requires the use of anti-anginal medication
* Ventricular arrhythmias except for benign premature ventricular contractions
* Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
* Conduction abnormality requiring a pacemaker
* Valvular disease with document compromise in cardiac function
* Symptomatic pericarditis
* Myocardial infarction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function
* History of documented congestive heart failure (New York Heart Association functional classification III-IV)
* Documented cardiomyopathy
* Patient has poorly controlled diabetes mellitus or steroid-induced diabetes mellitus
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol

  * Significant symptomatic deterioration of lung function; if clinically indicated, pulmonary function tests including measures of predicted lung volumes, diffusion capacity of the lung for carbon monoxide (DLCO), oxygen (O2) saturation at rest on room air should be considered to exclude pneumonitis or pulmonary infiltrates
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BJM120 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection); patients with unresolved diarrhea will be excluded as previously indicated; patients must be able to swallow capsules whole
* Patients who have been treated with any hematopoietic colony-stimulating growth factors (e.g., filgrastim [G-CSF], sargramostim [GM-CSF]) =< 2 weeks prior to starting study drug; erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to enrollment, may be continued
* Patients who are currently receiving treatment with medication with a known risk to prolong the QT interval or inducing Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug
* Patients receiving chronic treatment with steroids or another immunosuppressive agent; note: topical applications (e.g. rash), inhaled sprays (e.g. obstructive airway diseases), eye drops or local injections (e.g. intra-articular) are allowed; patients with previously treated brain metastases, who are on stable low dose corticosteroids treatment (e.g. dexamethasone 2 mg/day, prednisolone 10 mg/day) for at least 14 days before start of study treatment are eligible; premedication dexamethasone for pemetrexed is allowed
* Patients who are currently treated with drugs known to be strong inhibitors or inducers of isoenzyme cytochrome P450, family 3, subfamily A (CYP3A), and the treatment cannot be discontinued or switched to a different medication prior to starting study drug (please note that co-treatment with weak and moderate inhibitors and inducers of CYP3A is allowed)
* Herbal preparations/medication including but are not limited to St. John's wort, kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone [DHEA], yohimbe, saw palmetto, ginseng; patients should stop using these herbal medications 7 days prior to first dose of study drug
* Patients who have received systemic chemotherapy =< 4 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C) and prior to starting study drug toxicities must recover to a grade 1 before starting the trial
* Patients who have received any continuous or intermittent small molecule therapeutics (excluding monoclonal antibodies) =< 5 effective half lives prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who have received wide field radiotherapy =< 4 weeks or limited field radiation for palliation =< 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who have undergone major surgery =< 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who are currently taking therapeutic doses of warfarin sodium (Coumadin) or any other warfarin-derivative anticoagulant
* Women who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control; double barrier contraceptives must be used through the trial by both sexes; women of child-bearing potential, defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months), must have a negative serum pregnancy test =< 72 hours prior to initiating treatment

  * Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum follicle stimulating hormone (FSH) levels > 40 mIU/mL (for United States [US] only: and estradiol < 20 pg/mL) or have had surgical bilateral oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential
  * Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during treatment for 5 T1/2 (8 days) after stopping treatment and for additional 12 weeks (3 months in total after study drug discontinuation); the highly effective contraception is defined as either:
  * True abstinence: when this is in line with the preferred and usual lifestyle of the subject; periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago; in case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate); for female subjects on the study, the vasectomized male should be the sole partner for that patient
  * Use of a combination of any two of the following (a + b):

    * a) Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    * b) Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
  * Oral contraception, injected or implanted hormonal methods are not allowed
  * Fertile males, defined as all males physiologically capable of conceiving offspring, must use a condom during treatment, for 5 T1/2 (8 days) after stopping treatment and for an additional 12 weeks (3 months in total after study drug discontinuation) and should not father a child in this period
* Known diagnosis of human immunodeficiency virus (HIV) infection
* History of another malignancy within 3 years, except cured basal cell carcinoma of the skin or excised carcinoma in situ of the cervix
* Patient is unable or unwilling to abide by the study protocol or cooperate fully with the investigator
* Patient has acute viral hepatitis or a history of chronic or active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, (typically defined by elevated AST/ALT [persistent or intermittent], high HBV deoxyribonucleic acid [DNA] level hepatitis B virus surface protein antigen [HBsAg] positive, or high HCV ribonucleic acid [RNA] level) (testing not mandatory)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose, defined as the highest dose in which fewer than 33% of study participants experience a dose limiting toxicity (DLT), graded according to the National Cancer Institute (NCI) CTCAE version 4.0 | 21 days
Toxicity profile of PI3K inhibitor BKM120, assessed using NCI CTCAE version 4.0 | Up to 28 days after completion of study treatment
  Tables will be created to summarize all toxicities and side effects by dose, course, organ, and severity.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameters of PI3K inhibitor BKM120, carboplatin, and pemetrexed disodium in combination | Days 1 and 8 of course 1
  Means and 95% confidence intervals will be provided for the PK parameters.
Anti-tumor activity (complete response [CR] + partial response [PR]), assessed using RECIST | Up to 28 days after completion of study treatment
  Rates and associated 95% exact Clopper and Pearson binomial confidence limits will be estimated.
Disease control rate (CR + PR + stable disease [SD]), assessed using RECIST | Up to 28 days after completion of study treatment
  Rates and associated 95% exact Clopper and Pearson binomial confidence limits will be estimated.
Progression free survival | 6 months
  Rates and associated 95% exact Clopper and Pearson binomial confidence limits will be estimated.
Overall survival | 1 year
  Rates and associated 95% exact Clopper and Pearson binomial confidence limits will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Reckamp, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States